CLINICAL TRIAL: NCT06745661
Title: Investigating the Impact of RLRL on Alleviating Visual Fatigue in Presbyopic Population
Brief Title: Impact of Red Light Therapy on Alleviating Visual Fatigue in Presbyopes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSEARS20240916007
Record Dates: First submitted 2024-12-08; First posted 2024-12-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2024-12

CONDITIONS: Asthenopia; Visual Fatigue; Presbyopia
Keywords: asthenopia; visual fatigue; presbyopia; red light therapy
MeSH Terms: conditions — Asthenopia; Presbyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RLRL therapy group (Experimental): The experimental group will undergo repeated low-level red-light therapy (RLRL). The light power through a 4-mm pupil is 0.29 mW for the RLRL device.
  Interventions: Device: RLRL device
- Sham therapy group (Sham Comparator): The sham group will use a sham device, which operates at only 10% of the active RLRL device's power. The light power through a 4-mm pupil is 0.03 mW for the sham device.
  Interventions: Device: sham device

INTERVENTIONS:
Device: RLRL device — Each participant in the intervention group will be provided a repeated low-level red-light therapy (RLRL) device, which they are required to use twice daily for 3 minutes per session, with a minimum interval of 4 hours between sessions, 7 days a week for one month.
  Arms: RLRL therapy group
Device: sham device — Each participant in the sham group will be provided a sham therapy device, which they are required to use twice daily for 3 minutes per session, with a minimum interval of 4 hours between sessions, 7 days a week for one month.
  Arms: Sham therapy group

SUMMARY:
Visual fatigue, or asthenopia, occurs when visual demands exceed the capacity of the visual system, leading to various ocular discomfort and systemic symptoms. This condition can negatively affect personal activities, quality of life, and work productivity. Given the high prevalence of asthenopia in presbyopic population, finding effective methods to alleviate these symptoms is crucial. This study aims to evaluate the effects of repeated low-level red-light (RLRL) therapy on alleviating visual fatigue in individuals with presbyopia over a one-month period. Additionally, we will assess the potential benefits on accommodation function, cognition, and emotional effects of RLRL in this population.

Interested individuals will be invited to the PolyU Optometry Clinic to undergo an eligibility examination. An estimated sample size of 66 participants will be recruited. The inclusion criteria specify individuals aged 40 years or older who self-report visual fatigue symptoms and require near correction in daily life. Exclusion criteria include those with ocular disease, systemic diseases, illiteracy, or an afterimage duration longer than 6 minutes.

Eligible participants will be randomly assigned in a 1:1 ratio to either the intervention group or the control group. Each participant in the intervention group will be provided an RLRL therapy device, which they are required to use twice daily for 3 minutes per session, with a minimum interval of 4 hours between sessions, 7 days a week for one month. Participants in the control group will receive a sham device, following the same usage schedule. The study will evaluate changes in asthenopia questionnaire scores, CFF scores, other objective asthenopia indicators (i.e., eye movement, pupil parameters, and blink patterns), accommodation function, cognitive function, and emotional states at 2 weeks and 1 month compared to baseline. Statistical analysis will be conducted to explore evaluate within-subject changes over time and between-group differences in visual fatigue metrics, accommodation metrics, cognitive metrics, and emotional metrics.

The findings will contribute to evaluating the effectiveness of RLRL therapy in reducing asthenopia and presbyopia symptoms, as well as its impact on cognitive function and emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged over 40 years old.
* Self-reported visual fatigue symptoms.
* Distance best-corrected visual acuity (BCVA) of 0.5 LogMAR or better, and near visual acuity worse than N8 (20/50) at 40 cm with the subject's habitual distance correction.
* Require near correction in daily life.
* No light therapy received in the past six months.
* Giving informed written consent.

Exclusion Criteria:

* Presence of diseases that can cause eye pain or headaches, such as strabismus, glaucoma, ocular trauma, conjunctivitis, migraines, keratitis, iridocyclitis, or other self-reported diseases.
* Systemic diseases (e.g., epilepsy, photosensitivity, seizure) or illiteracy.
* Afterimage time longer than 6 minutes.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
change in the asthenopia questionnaire scores | at 2 weeks and 1 month compared to baseline
  The primary outcome is the change in the asthenopia questionnaire scores at 2 weeks and 1 month compared to baseline. These scores will be derived from the Computer Vision Syndrome Questionnaire (CVS-Q), a widely recognized tool for assessing subjective symptoms of asthenopia. The CVS-Q ranges from 0 (no symptoms) to 32 (most severe), with higher scores indicating worse symptoms (negative change = improvement)

SECONDARY OUTCOMES:
Change in critical flicker fusion frequency (CFF) | at 2 weeks and 1 month compared to baseline
  •Change in CFF at 2 weeks and 1 month compared to baseline.
Change in eye movement | at 2 weeks and 1 month compared to baseline
  •Change in eye movement at 2 weeks and 1 month compared to baseline.
Change in pupil parameters | at 2 weeks and 1 month compared to baseline
  •Change in pupil parameters at 2 weeks and 1 month compared to baseline.
Change in blink patterns | at 2 weeks and 1 month compared to baseline
  •Change in blink patterns at 2 weeks and 1 month compared to baseline.
Change in accommodation function | at 2 weeks and 1 month compared to baseline
  •Change in accommodation function at 2 weeks and 1 month compared to baseline.
Change in self-reported emotional states | at 2 weeks and 1 month compared to baseline
  Change in self-reported emotional states, assessed by the Positive and Negative Affect Schedule (PANAS-X) at 2 weeks and 1 month compared to baseline. The scores are divided into positive scores and negative scores. Items are rated for the past week on a 5-point scale. The Positive Affect subscale (items 1,3,5,9,10,12,14,16,17,19) and Negative Affect subscale (items 2,4,6,7,8,11,13,15,18,20) each total 10-50 points.
  Positive Affect Score: Higher scores indicate higher levels of positive affect. Negative Affect Score: Lower scores indicate lower levels of negative affect.
Change in electroencephalogram (EEG) | at 2 weeks and 1 month compared to baseline
  •Change EEG at 2 weeks and 1 month compared to baseline.
Change in cognitive questionnaire | at 2 weeks and 1 month compared to baseline
  •Change in cognitive questionnaire, measured by the Montreal Cognitive Assessment Scale (MoCA) at 2 weeks and 1 month compared to baseline. Total score 0-30; higher scores indicate better cognitive function.
Change in near activity visual questionnaire | at 2 weeks and 1 month compared to baseline
  Change in near activity visual questionnaire (NAVQ) score at 2 weeks and 1 month compared to baseline. Scores are reported on the Rasch-transformed 0-100 scale, with higher scores indicating worse near-vision function (decreases = improvement).

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytchnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
According to the relevant agreement, all parties involved must keep study data confidential throughout the study process.